CLINICAL TRIAL: NCT03282955
Title: A Randomized, Controlled, Double-blind, Multicenter Clinical Trial on Home Parenteral Nutrition Using an Omega-3 Fatty Acid Enriched MCT/LCT Lipid Emulsion
Brief Title: The HOME Study (HPN With OMEGA-3)
Acronym: HOME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC-G-H-1403
Record Dates: First submitted 2017-08-10; First posted 2017-09-14 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Patients Requiring Home Parenteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lipidem (Experimental): i.v. lipid emulsion containing fractionated fish oil (n-3 fatty acid triglycerides)
  Interventions: Drug: Lipidem
- Lipofundin MCT (Active Comparator): i.v. lipid emulsion
  Interventions: Drug: Lipofundin MCT 20%

INTERVENTIONS:
Drug: Lipidem — Lipoplus i.v. lipid emulsion for parenteral nutrition
  Arms: Lipidem
Drug: Lipofundin MCT 20% — Lipofundin MCT 20% i.v. lipid emulsion for parenteral nutrition
  Arms: Lipofundin MCT

SUMMARY:
The aim of the trial is to investigate safety and tolerability of an Omega-3-FA-enriched lipid emulsion in adult patients with chronic intestinal failure in need of long-term HPN. It is aimed to show non-inferiority of the lipid emulsion Lipidem (investigational test product) in comparison to the lipid emulsion Lipofundin MCT (investigational reference product) with regard to liver function.

ELIGIBILITY:
Inclusion:

* Signed informed consent available
* Male or female patients ≥ 18 years of age
* Patients with chronic intestinal failure receiving HPN including lipids in whom the parenteral macronutrients have not been changed by more than 10% for at least 3 months
* Patients receiving ≥ 3.0 g lipids/kg body weight per week

Exclusion:

* Persistent high total bilirubin values in medical history of last 6 months (> 40µmol/l)
* Patients in whom PN was interrupted for longer than 4 continuous weeks in the preceding 6 months
* Patients with history of cancer and anti-cancer treatment within the last 2 years
* Hypersensitivity to egg, fish, peanut or soya-bean protein or to any of the active substances or excipients
* Patients treated in the past or currently with Teduglutide
* Contraindications to investigational products (if available from medical records) including:

  * Severe hyperlipidemia, including severe hypertriglyceridaemia (≥1000 mg/dl or 11.4 mmol/l)
  * Severe coagulopathy
  * Intrahepatic cholestasis
  * Severe hepatic insufficiency
  * Severe renal insufficiency in absence of renal replacement therapy
  * Acute thromboembolic events
  * Fat embolism
  * Aggravating haemorrhagic diatheses
  * Metabolic acidosis
* General contraindications to parenteral nutrition (if available from medical records) including:

  * Unstable circulatory status with vital threat (states of collapse and shock)
  * Acute phase of cardiac infarction or stroke
  * Unstable metabolic conditions (e.g. decompensated diabetes mellitus, severe sepsis, coma of unknown origin)
  * Inadequate cellular oxygen supply
  * Disturbances of the electrolyte and fluid balance (e.g. hypokalaemia and hypotonic dehydration)
  * Acute pulmonary edema
  * Decompensated cardiac insufficiency
* Positive test for HIV, Hepatitis B or C (from medical history)
* Known or suspected drug or alcohol abuse
* Patients who are unwilling or mentally and/or physically unable to adhere to study procedures
* Participation in another interventional clinical trial in parallel or within three months prior to the start of this clinical trial
* Any medical condition that in the opinion of the investigator might put the subject at risk or interfere with patients participation For women with childbearing potential (i.e. females who are not chemically or surgically sterile or females who are not post-menopausal)
* Women of childbearing potential tested positive on standard pregnancy test (urine dipstick)
* Lactation
* Women of childbearing potential who do not agree to apply adequate contraception
* Persons of legal age who are the subject of a legal protection measure or who are unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- France (2):
  - Hôpital Archet 2 - Unité de support nutritionnel, Nice
  - Hospices Civiles de Lyon - Centre hospitalier Lyon Sud, Pierre-Bénite
- Department of Medical and Surgical Science, University of Bologna, Center for Chronic Intestinal Failure, Department of Digestive System, St. Orsola-Malpighi Hospital, Bologna, Italy
- Radboud university medical center, Nijmegen, Netherlands
- Poland (3):
  - Wojewódzkim Specjalistycznym Szpitalem im. M. Pirogowa w Łodzi , Oddział Chirurgii Ogólnej i Naczyniowej, Lodz
  - Stanley Dudrick's Memorial Hospital, Skawina
  - Samodzielny Publiczny Szpital Kliniczny, im. prof. dr W. Orlowskiego, Centrum Medycznego Ksztalcenia Podyplomowego, Oddzial Kliniczny Zywienia i Chirurgii, Warsaw
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University College Hospital London, London

REFERENCES:
- [Derived] Klek S, Chambrier C, Szczepanek K, Kunecki M, Sobocki J, Wanten G, Pironi L, Schneider SM, Rahman F, Cooper SC, Calder PC, Gabe S, Forbes A. Safe and well-tolerated long-term parenteral nutrition regimen: Omega-3-fatty-acid-enriched medium chained/ long chained triglycerides emulsion. Clin Nutr. 2024 Dec;43(12):415-424. doi: 10.1016/j.clnu.2024.11.007. Epub 2024 Nov 7. PMID 39581180
- [Derived] Klek S, Chambrier C, Cooper SC, Gabe S, Kunecki M, Pironi L, Rahman F, Sobocki J, Szczepanek K, Wanten G, Lincke N, Glotzbach B, Forbes A. Home parenteral nutrition with an omega-3-fatty-acid-enriched MCT/LCT lipid emulsion in patients with chronic intestinal failure (the HOME study): study protocol for a randomized, controlled, multicenter, international clinical trial. Trials. 2019 Dec 30;20(1):808. doi: 10.1186/s13063-019-3994-z. PMID 31888740

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lipidem | Lipofundin MCT
Started | 40 | 34
Completed | 35 | 30
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Population: 74 patients were enrolled for the study. However, 2 patients dropped out before any further intervention. Therefor these 2 patients were not included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lipidem | Lipofundin MCT | Total
Number analyzed (Participants) | 38 | 34 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.13 (15.82) | 52.44 (15.50) | 51.22 (15.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 24 | 40
  Male | 22 | 10 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35 | 31 | 66
  Black or African American | 1 | 0 | 1
  Native Hawaiian/Other Pacific | 0 | 1 | 1
  Missing | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Netherlands | 4 | 3 | 7
  Poland | 20 | 16 | 36
  Italy | 2 | 3 | 5
  United Kingdom | 2 | 1 | 3
  France | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change of Liver Function Parameters From Baseline to Visit 2
Description: Changes will be expressed as the sum of the N(0.1)- transformed differences of bilirubin, ALT and AST (from Baseline to Visit 2), i.e. for all three parameters each change of the value is subtracted by the mean change of the respective parameter. This difference is divided by the standard deviation of the change, which results in a unitless normalised value. All values for the 3 liver parameters (bilirubin, ALT and AST) will be added. The final sum reflects the change of liver function parameters.
Time Frame: 8 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: normalized sum- no unit
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 36 | 31
normalized sum- no unit | 0.0606 (3.0876) | -0.0703 (1.8063)
Statistical Analysis 1: Comparison: Lipidem vs Lipofundin MCT; Test type: Non-Inferiority — Non-inferiority margin= 1.151; p = 0.025, t-test, 1 sided

2. Secondary Outcome: Bilirubin
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 36 | 31
µmol/L | 0.36 (3.34) | 0.04 (3.26)

3. Secondary Outcome: Alanine Transaminase (ALT)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: µkat/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 36 | 31
µkat/L | 0.06 (0.60) | 0.01 (0.25)

4. Secondary Outcome: Aspartate Transaminase (AST)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: µkat/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 36 | 31
µkat/L | -0.03 (0.38) | -0.00 (0.21)

5. Secondary Outcome: AST/ALT Ratio
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 34 | 31
Ratio | 0.53 (1.00) | 0.89 (2.52)

6. Secondary Outcome: Alkaline Phosphatase (ALP)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: µkat/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 34 | 30
µkat/L | 0.13 (0.66) | -0.15 (1.46)

7. Secondary Outcome: Gamma-glutamyl Transpeptidase (GGT)
Description: Change from baseline
Time Frame: 8 weeks
Population: Safety Set
Measure: Mean (Standard Deviation); unit: µkat/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 35 | 30
µkat/L | 0.02 (0.38) | -0.11 (1.64)

8. Secondary Outcome: White Blood Cells (WBCs)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 34 | 31
10^9 cells/L | 0.45 (1.42) | 0.19 (1.39)

9. Secondary Outcome: Red Blood Cells (RBCs)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 34 | 31
10^12 cells/L | -0.02 (0.28) | -0.10 (0.28)

10. Secondary Outcome: Hemoglobin (Hb)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: g/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 34 | 31
g/L | 0.52 (8.82) | -1.75 (8.22)

11. Secondary Outcome: Platelets
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 34 | 31
10^9 cells/L | 3.06 (41.11) | 6.90 (50.33)

12. Secondary Outcome: International Normalized Ratio (INR) (if Not Possible Prothrombin Time [PT = Quick-value] is Accepted)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 27 | 25
Ratio | -0.01 (0.25) | -0.16 (0.71)

13. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 25 | 19
seconds | 0.02 (3.85) | 0.97 (7.69)

14. Secondary Outcome: Hematocrit (Hct)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 34 | 31
L/L | -0.00 (0.03) | -0.01 (0.03)

15. Secondary Outcome: Blood Glucose
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 32 | 31
mmol/L | 0.43 (0.94) | -0.14 (1.33)

16. Secondary Outcome: Sodium
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 35 | 31
mmol/L | 0.18 (2.67) | -0.58 (2.74)

17. Secondary Outcome: Chloride
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 35 | 31
mmol/L | -0.19 (3.33) | -0.15 (4.08)

18. Secondary Outcome: Potassium
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 35 | 31
mmol/L | 0.06 (0.37) | 0.01 (0.46)

19. Secondary Outcome: Calcium
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 35 | 31
mmol/L | -0.01 (0.15) | -0.01 (0.10)

20. Secondary Outcome: Magnesium
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 35 | 30
mmol/L | 0.00 (0.09) | -0.00 (0.06)

21. Secondary Outcome: Phosphate
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 34 | 30
mmol/L | -0.02 (0.18) | -0.00 (0.16)

22. Secondary Outcome: Serum Creatinine
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 35 | 31
µmol/L | 3.87 (32.42) | 0.43 (9.23)

23. Secondary Outcome: Triglycerides
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 36 | 30
mmol/L | 0.10 (0.55) | 0.19 (0.68)

24. Secondary Outcome: Cholesterol
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 36 | 30
mmol/L | 0.01 (0.39) | 0.02 (0.71)

25. Secondary Outcome: High-density Lipoprotein (HDL)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 36 | 30
mmol/L | -0.12 (0.19) | 0.03 (0.23)

26. Secondary Outcome: Low-density Lipoprotein (LDL)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 36 | 30
mmol/L | 0.07 (0.33) | -0.08 (0.76)

27. Secondary Outcome: C-reactive Protein (CRP)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 35 | 30
nmol/L | 37.16 (160.03) | -24.65 (209.18)

28. Secondary Outcome: α-Tocopherol/Vitamin E (Facultative if Routinely Assessed)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: µmol/L]
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 4 | 5
µmol/L] | -3.00 (6.60) | -1.94 (10.99)

29. Secondary Outcome: Triene:Tetraene Ratio in Plasma, Reduction From Baseline
Description: Derived from fatty acid pattern in plasma
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 34 | 27
Ratio | 0.011 (0.024) | 0.008 (0.028)

30. Secondary Outcome: Adverse Events
Description: Number of adverse events (including serious adverse events)
Time Frame: 8 weeks
Measure: Number; unit: Adverse events
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 38 | 34
Adverse events | 31 | 25

31. Secondary Outcome: BMI
Description: Body mass index Change from baseline
Time Frame: 8 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 36 | 31
kg/m^2 | 0.4 (0.7) | 0.2 (0.7)

32. Secondary Outcome: Prothrombin Time (PT)
Description: Change from baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Lipidem | Lipofundin MCT
Number analyzed (Participants) | 6 | 3
s | -0.8 (1.15) | 1.27 (5.16)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Lipidem | Lipofundin MCT
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/34
Serious Adverse Events (participants affected / at risk) | 5/40 | 3/34
Other Adverse Events (participants affected / at risk) | 15/40 | 12/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipidem (N=40) | Lipofundin MCT (N=34)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 0 (0)
Dermo-hypodermitis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Device dislocatioin (Product Issues) | 0 (0) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipidem (N=40) | Lipofundin MCT (N=34)
White blood cell (Investigations) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine Aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Asparte Aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Dyspnoe exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Deep vein thrombosis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Device infusion issue (Product Issues) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In order to ensure that the Sponsor will be able to make comments and suggestions where pertinent, material for public dissemination will be submitted to the Sponsor for review at least sixty (60) days (or longer if specified elsewhere) prior to submission for publication, public dissemination, or review by a publication committee.

The PI agrees that all reasonable comments made by the Sponsor in relation to a proposed publication will be incorporated into the publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT03282955/Prot_SAP_000.pdf